CLINICAL TRIAL: NCT07200583
Title: Efficacy and Safety of Protein A Immunoadsorption-Based Desensitization in Highly Sensitized Haploidentical Hematopoietic Stem Cell Transplantation: A Single-Center Retrospective Study
Brief Title: Protein A Immunoadsorption in Highly Sensitized Haplo-HSCT Patients
Acronym: PAIA-Haplo
Status: Completed | Type: Observational
Sponsor: Ting YANG (Other)
Responsible Party: Sponsor-Investigator, Ting YANG, Prof., Fujian Medical University
Organization: Fujian Medical University (Other)
Other Study IDs: DSA-PAIA-01
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hematologic Malignancies; Hematologic Disorders; Allogeneic Hematopoietic Stem Cell Transplantation (HSCT); Graft Failure
Keywords: Haploidentical HSCT; Donor-specific anti-HLA antibodies (DSA); Protein A immunoadsorption; Desensitization therapy; Primary graft failure; Poor graft function; Engraftment; Rituximab; Bortezomib
MeSH Terms: conditions — Hematologic Neoplasms; Hematologic Diseases | interventions — Rituximab; Bortezomib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Desensitization Group: Highly sensitized haplo-HSCT patients who received protein A immunoadsorption-based desensitization therapy.
  Interventions: Procedure: Protein A immunoadsorption; Drug: Rituximab (optional, in some patients); Drug: Bortezomib (optional, in some patients)

INTERVENTIONS:
Procedure: Protein A immunoadsorption — Extracorporeal therapy performed prior to haploidentical HSCT to remove donor-specific anti-HLA antibodies (DSA)
Drug: Rituximab (optional, in some patients) — Anti-CD20 monoclonal antibody occasionally combined with immunoadsorption as part of desensitization strategy
Drug: Bortezomib (optional, in some patients) — Proteasome inhibitor occasionally used in combination with desensitization therapy.

SUMMARY:
This study reviews patients who received haploidentical hematopoietic stem cell transplantation (haplo-HSCT). Some patients develop donor-specific antibodies (DSA), which can block engraftment and cause transplant failure. Before transplant, a treatment called protein A immunoadsorption (a blood purification method to remove antibodies) was used, sometimes with additional medications.

The study aims to see whether this approach lowers antibody levels, increases the chance of successful engraftment, reduces complications such as infections or graft failure, and improves short-term survival. The results may help guide safer and more effective transplants for highly sensitized patients.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) is an effective, and often the only curative, treatment for many malignant and non-malignant hematologic diseases. Haploidentical HSCT (haplo-HSCT) has become a widely available option, but the presence of donor-specific anti-HLA antibodies (DSA) in recipients significantly increases the risk of graft rejection and primary graft failure. High DSA levels, particularly with mean fluorescence intensity (MFI) ≥5000, have been shown to result in substantially higher rates of engraftment failure compared with patients without DSA.

To address this problem, desensitization strategies are needed. Protein A immunoadsorption is an extracorporeal therapy that selectively removes antibodies from the blood and may reduce the risk of graft failure. In this single-center, retrospective study, we will evaluate the efficacy and safety of protein A immunoadsorption-based desensitization, sometimes combined with agents such as rituximab or bortezomib, in highly sensitized haplo-HSCT patients.

The primary outcome is hematopoietic engraftment success rate. Secondary outcomes include changes in DSA levels (MFI reduction, clearance, or negativity), incidence of major transplant-related complications (primary graft failure, poor graft function, severe infections, acute graft-versus-host disease), and survival outcomes (overall survival and disease-free survival at 100 days and 1 year). Risk factor analysis will also be performed to identify predictors of engraftment failure or poor survival.

Because this is a retrospective observational study, no additional interventions will be introduced, and all data will be collected from medical records. This research is expected to provide real-world evidence to optimize desensitization strategies and improve clinical outcomes in highly sensitized haplo-HSCT recipients.

ELIGIBILITY:
Inclusion Criteria:

Patients who received haploidentical allogeneic hematopoietic stem cell transplantation (haplo-HSCT) from a related donor (≥5/10 HLA match).

Presence of donor-specific anti-HLA antibodies (DSA) before transplantation, with mean fluorescence intensity (MFI) above the positive threshold.

Underwent desensitization therapy mainly based on protein A immunoadsorption (with or without additional agents such as rituximab or bortezomib), with complete treatment records.

Successfully completed transplantation at the study center and had at least 100 days of follow-up.

Exclusion Criteria:

Missing critical data (e.g., incomplete DSA results, desensitization details, or follow-up outcomes).

Inadequate follow-up (patients lost to follow-up or transferred to another hospital without accessible records).

Patients who did not complete desensitization or did not undergo HSCT infusion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Highly sensitized patients with donor-specific anti-HLA antibodies (DSA positive) who underwent haploidentical hematopoietic stem cell transplantation at the First Affiliated Hospital of Fujian Medical University and received protein A immunoadsorption-based desensitization therapy prior to transplant.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2025-05-31 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Hematopoietic engraftment success rate | Within 28 days after transplantation
  Proportion of patients achieving engraftment after haploidentical HSCT, defined as:
  Neutrophil recovery ≥0.5 × 10^9/L for 3 consecutive days; Platelet recovery ≥20 × 10^9/L without transfusion for 3 consecutive days

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian 350001, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No